CLINICAL TRIAL: NCT00835952
Title: Phase 1, Open-label Study of the Safety, Tolerability, and Histological Effect of Single Doses of ATX-101 (Sodium Deoxycholate for Injection) Administered in Abdominal Fat in Subjects Undergoing Abdominoplasty
Brief Title: ATX-101 Abdominoplasty
Acronym: ATX-101-08-10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Director, Clinical Affairs, Kythera Biopharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ATX-101-08-10
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Characteristics of Subcutaneous Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATX-101 (Experimental)
  Interventions: Drug: ATX-101

INTERVENTIONS:
Drug: ATX-101 — ATX-101 single doses

SUMMARY:
Histopathological study of abdominal fat excised from subjects undergoing abdominoplasty

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects undergoing planned abdominoplasty

Exclusion Criteria:

* History of interventions in the abdominal area

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory test results, physical examinations | 1 - 28 days

SECONDARY OUTCOMES:
Histopathology | 1 - 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, M.D., Ph.D., Study Director — Kythera Biopharmaceuticals, Inc.
Locations (2):
- United States (2):
  - San Francisco, California
  - Santa Monica, California